CLINICAL TRIAL: NCT02401438
Title: Accuracy of 5D LB Ultrasound in Predicting Birth Weight of Preterm Fetuses : A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, professor, Ain Shams University
Other Study IDs: m2494
Record Dates: First submitted 2015-03-19; First posted 2015-03-27 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pregnant women with preterm delivery: 5D LB and 2D ultrasounds will be done to pregnant women between 28 and 34 weeks planned for termination of pregnancy for obstetric or medical causes.
  Interventions: Other: 5D ultrasound; Other: 2D ultrasound

INTERVENTIONS:
Other: 5D ultrasound
Other: 2D ultrasound

SUMMARY:
5D and 2D ultrasound will be done for pregnant women within 72hours before preterm delivery to determine estimated fetal weight by ultrasound. The estimated fetal weight by 5D and 2D ultrasound will be compared to the actual birth weight to determine accuracy of 5D ultrasound in predicting actual birth weight .

ELIGIBILITY:
Inclusion Criteria:

* 28 to 34 weeks
* preterm termination of pregnancy
* singleton pregnancy
* any obstetric or medical cause for termination of pregnancy

Exclusion Criteria:

* IUFD
* multiple pregnancy
* congenital anomalies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women between 28 and 34 weeks scheduled for termination of pregnancy due to medical or obstetric cause
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Accuracy of 5D ultrasound in predicting actual birth weight in preterm fetuses | 72hours
  Sensitivity specificity positive predictive value and negative predictive values will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt